CLINICAL TRIAL: NCT00039312
Title: Multi-Institutional Prospective Cohort Study For The Comparison Of Different Primary Screening Strategies For The Detection Of Cervical Neoplasia
Brief Title: Comparison of Screening Tests in Detecting Cervical Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Purpose: Screening
Other Study IDs: 99-10-034; UCLA-9910034; NCI-G02-2076
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Cervical Cancer
Keywords: cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papanicolaou Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Papanicolaou test
Other: cytology specimen collection procedure
Procedure: annual screening
Procedure: colposcopic biopsy
Procedure: comparison of screening methods

SUMMARY:
RATIONALE: Screening tests may help doctors detect abnormal cells in the cervix early and plan effective treatment.

PURPOSE: Screening trial to compare different types of screening tests used to detect cervical neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the sensitivity and specificity of primary screening strategies for the detection of cervical intraepithelial or invasive neoplasia.
* Compare the positive and negative predictive values of these strategies.

OUTLINE: This is a multicenter study. Patients are stratified according to the reason for the visit (general gynecological screening vs colposcopy referral).

* Stratum 1 (general gynecological screening): Patients undergo Pap smear, visual inspection aided by acetic acid (VIA), a colposcopy, and finally a visual inspection aided by toluidine blue (VIT) followed by an acetic acid wash. A biopsy may be performed at this initial visit. Within 2-3 weeks, patients are notified of results.
* Stratum 2 (colposcopy referral): Patients undergo Pap smear, VIA, colposcopy, VIT, and possible biopsy as in stratum 1. During the same visit, patients receive histologic evaluation and treatment with See-and-Treat loop electrosurgical excision procedure and/or endocervical curettage.

PROJECTED ACCRUAL: A total of 600-1,000 patients (300-500 per stratum) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria::

* History of cervical neoplasia
* Presenting for a well-woman visit, annual Pap smear, or family planning

  * Other gynecological or non-gynecological complaints allowed OR
* Referred for colposcopy secondary to an abnormal Pap smear
* Planned screening for cervical cancer
* Over 18 years of age
* Prior laser surgery, cryotherapy, or conization or loop electrosurgical excision procedure for cervical neoplasia allowed

Exclusion Criteria:

* bleeding diathesis
* pregnant
* prior hysterectomy
* concurrent anticoagulants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1999-12; Primary Completion 2003-08 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Holschneider, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States